CLINICAL TRIAL: NCT01077245
Title: A Phase 2 Study to Evaluate the Safety and Potential Efficacy of Clostridium Butyricum MIYAIRI 588 Strain (MIYA-BM Fine Granules) for the Prevention of Recurrent Clostridium Difficile Infections
Brief Title: Safety and Clinical Effectiveness of Oral Probiotic MIYA-BM to Prevent Recurrent Clostridium Difficile Infections
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Osel, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-001
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Clostridium Infections; Gram-Positive Bacterial Infections; Bacterial Infections; Anti-Infective Agents; Clostridium butyricum; Metronidazole; Vancomycin; Gastrointestinal Diseases; Physiological Effects of Drugs; Colonic Diseases; Enterocolitis, Pseudomembranous; Intestinal Diseases; Enterocolitis; Pharmacologic Actions; Digestive System Diseases; Therapeutic Uses; Gastroenteritis; Colitis; Diarrhea; Probiotics; Gastrointestinal Agents
MeSH Terms: conditions — Clostridium Infections; Gram-Positive Bacterial Infections; Bacterial Infections; Gastrointestinal Diseases; Colonic Diseases; Enterocolitis, Pseudomembranous; Intestinal Diseases; Enterocolitis; Digestive System Diseases; Gastroenteritis; Colitis; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIYA-BM (Experimental): MIYA-BM Fine Granules (CBM588)
  Interventions: Drug: MIYA-BM Fine Granules (CBM588)
- Placebo (Placebo Comparator): Placebo Fine Granules (without CBM588)
  Interventions: Drug: Placebo Fine Granules (without CBM588)

INTERVENTIONS:
Drug: MIYA-BM Fine Granules (CBM588) — MIYA-BM Fine Granules (CBM588)
  Arms: MIYA-BM
Drug: Placebo Fine Granules (without CBM588) — Placebo Fine Granules (without CBM588)
  Arms: Placebo

SUMMARY:
Patients with confirmed C. difficile infection (CDI) who meet eligibility requirements will be invited to participate. All study patients must receive treatment for CDI with metronidazole or vancomycin. Enrolled patients will be randomized in a 1:1 ratio to receive MIYA-BM Fines Granules [Clostridium butyricum MIYAIRI 588 Strain (CBM588)] or a placebo orally twice a day for 42 days. Patients will be evaluated for safety and clinical outcomes through Day 180. Occurrence of adverse events (AEs), diarrhea history, and concomitant medications will be evaluated at scheduled study visits and telephone contacts.

DETAILED DESCRIPTION:
This study is a Phase 2 blinded, placebo-controlled, randomized clinical trial of an oral probiotic product, MIYA-BM Fine Granules [Clostridium butyricum MIYAIRI 588 Strain (CBM588)], in patients diagnosed with CDI and treated with metronidazole or vancomycin. Two hundred patients who meet all eligibility criteria will be randomized in a 1:1 fashion to receive either MIYA-BM (2g/dose) or placebo orally twice daily for 42 days. After randomization, all patients will be followed for a total of 180 days (6 months) for safety and recurrent CDI. If initially hospitalized, patients will be followed daily for diarrhea history, collection of concomitant medications and AEs, and monitored for their response to treatment. Patients will be followed through clinic visits and safety telephone calls. All patients will be given a Diary Card to report AEs, diarrhea history, and concomitant medications on a daily basis. If patients have signs or symptoms of CDI following resolution of the initial episode, they will be instructed to return to the clinic as soon as possible for evaluation of recurrent CDI. If a patient is diagnosed with recurrent CDI, they will discontinue study treatment (MIYA-BM or placebo) and be treated and followed according to the institution's standard of care for recurrent CDI.

ELIGIBILITY:
Inclusion Criteria:

* Adult of either gender, aged 18-80 years old inclusive
* Meets the case definition of CDI - recent history of diarrhea with presence of C. difficile toxin or pseudomembranous colitis; and no other known etiology of diarrhea (e.g. other enteric pathogen, other intestinal disease)
* CDI treated with metronidazole or vancomycin
* If female and of reproductive potential, subject must not be pregnant (negative pregnancy test at time of screening) or breast-feeding, and currently using a reliable method of birth control

Exclusion Criteria:

* Has other known etiology of diarrhea (e.g. other enteric pathogen, other intestinal disease)
* Has a history of acute pancreatitis within the last 3 months
* Has a history of chronic intestinal disease (e.g. Crohn's disease, ulcerative colitis)
* Is unable to complete a daily study diary (mental incapacity, head trauma, etc.)
* Has presence of toxic megacolon or ileus
* Has presence of colostomy, naso-gastric tube, or indwelling central line
* Has history of abdominal surgery within the previous 3 months (from time of enrollment)
* Has recent history of other investigational drug use within 30 days of enrollment visit
* Has planned investigational drug use while participating in this study
* Is known to have HIV infection or AIDS or other immunosuppressive disease
* Has taken systemic immunosuppressive drugs within 60 days of enrollment
* Is currently taking or is planning to use an oral probiotic, other than yogurt, during the study
* Has a known allergy to any component of MIYA-BM Fine Granules or placebo
* Is unavailable for follow-up visits
* At enrollment, has any social or medical condition, or psychiatric illness that, in the opinion of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of the study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety of MIYA-BM | 180 days
  Evaluation of the safety of MIYA-BM compared to placebo in patients with CDI who are treated with metronidazole or vancomycin by comparing the adverse events (AEs) and serious adverse events (SAEs) in the MIYA-BM and placebo groups, as well as observed and self-reported clinical signs and symptoms, physical findings, and laboratory measurements.

SECONDARY OUTCOMES:
Efficacy of MIYA-BM | 60 days
  Evaluation of the potential efficacy of MIYA-BM compared to placebo in the prevention of recurrent CDI as determined by the proportion of subjects with recurrent CDI and time to recurrence of the first CDI after initiation of MIYA-BM or placebo treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne V. McFarland, Ph.D., Principal Investigator — VA Puget Sound Health Care System